CLINICAL TRIAL: NCT05364970
Title: Immersive Virtual Reality in the Rehabilitation of Peripheral Injuries
Brief Title: IVR in Motor Rehabilitation
Acronym: IVR_MOT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: HastaFisio - Fisioterapia e Medicina dello Sport (Unknown)
Responsible Party: Principal Investigator, Lorenzo Pia, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1234
Record Dates: First submitted 2022-04-26; First posted 2022-05-06 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Knee Injuries
Keywords: Knee reconstruction; Immersive virtual reality; Full body illusion; Motor rehabilitation
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR_1PP (Experimental): Virtual training with an avatar observed from the first-person perspective
  Interventions: Combination Product: VR_Training_1PP
- VR_3PP (Active Comparator): Virtual training with an avatar observed from the third-person perspective
  Interventions: Combination Product: VR_Training_3PP
- NO_VR (No Intervention): No VR training administered

INTERVENTIONS:
Combination Product: VR_Training_1PP — Immersive VR scenario of physical training with avatar embodiment
  Arms: VR_1PP
Combination Product: VR_Training_3PP — Immersive VR scenario of physical training without avatar embodiment
  Arms: VR_3PP

SUMMARY:
The present project on sport rehabilitation aims at validating a rehabilitation protocol in immersive virtual reality (IVR) for restoring motor functions following peripheral injuries of the lower limbs. Sport injuries are related to direct and indirect costs and, in many cases, cause an interruption of motor activity for prolonged periods. Sport physiotherapy aims at recovering the motor functionality in order to guarantee the fastest possible return to sport. It employs plasticity and compensatory mechanisms within the injured motor system. However, being primarily based on the execution of movements that can be largely compromised, the treatment might be intrinsically complicated.

It has been suggested that the motor system can be activated by observing one's own body perform the movements, without any actual movement execution. By using multisensory integration and sense of presence in IVR, it is possible to create an illusory experience that a moving virtual body (avatar) temporarily becomes one's own moving body. Moreover, this experience activates the motor system similarly to the activation from one's own actual movements. Based on these considerations, the present study hypothesizes that observation of one's own virtual body, without any movement execution, might activate the motor system to the extent of significantly improving functional recovery.

The randomized clinical trial will recruit participants that underwent knee surgery and are in the first phase of the rehabilitation period (starting within two weeks after the surgery). Together with the traditional training protocol (4-6 weeks) participants will be administered a training in IVR that will include a virtual avatar performing a series of standard lower limb rehabilitation exercises. Participants will be randomly assigned to the experimental group (avatar observed from the first-person perspective, i.e., perceived as one's own body), the active control group (avatar observed from the third-person perspective, i.e., perceived as another person's body) and the group with no intervention. Before, at midpoint and after intervention, a standard battery of tests will be administered to evaluate the state of the motor system), as well as measures of embodiment for controlling the efficacy of the virtual scenario. The hypothesis is that the experimental group will show greater improvement of the motor functionality compared to the two control groups.

DETAILED DESCRIPTION:
BACKGROUND Sport injuries are an important obstacle both for sport performance and for maintaining a healthy lifestyle that implies continuous and regular physical activity. In Italy, each year there are approximately 300.000 admissions to the ER among 20 millions of people practicing sports.

As regards competitive sport, dense competition schedules, fast-paced rhythms and growing pressure experienced by athletes determine the increasing frequency of injuries. Injuries result in periods of refrain from competitions and affects athletes' psycho-physical balance. For these reasons, sport injuries have significant direct and indirect costs and physiotherapy aims to recover motor function to guarantee the fastest and safest return to sport.

Any form of motor rehabilitation, both in cases of damage to the central nervous system and those related to peripheral problems (as in the majority of sport injuries), is based on the concepts of plasticity and compensation. In other words, the possibility of recovery implies that the system can reorganize itself. In practical terms, rehabilitation science in its current form attempts to directly promote active and repetitive exercise of the damaged (motor) system. This logic, i.e., the process that is primarily based on action execution, has a major intrinsic limit that poses an obstacle for the treatment: it works directly with the motor functioning that is, however, compromised, even to a severe extent. However, it has been recently suggested that the motor system can be activated by simply observing one's own body perform the movements, without any actual movement execution. In line with that, and taking advantage of the multisensory nature and the sense of presence and embodiment that Immersive virtual reality (IVR) provides, it has been shown that it is possible to create an illusory experience that a moving virtual body (avatar) temporarily became one's own moving body (so-called embodiment. Moreover, this experience activates the motor system in a way similar to the activation from one's own actual movements. Therefore, in such conditions, the (illusory) movements of the embodied virtual body are integrated in the participant's motor system.

Based on these theoretical considerations, the present project proposes to employ the IVR to test a possible drastic change to the rehabilitation approach that would bypass/limit the problem of the (deficient) motor execution. The main hypothesis is that simple observation of a moving virtual body, which is perceived as one's own, would allow accessing the motor system to the extent of promoting the functional recovery. In other words, the aim is to access the motor functioning through the (intact) somatosensory system, rather than through the (damaged) motor one. In addition, such a procedure provides the possibility to perform at least a part of the treatment remotely.

AIMS

The present research project on sport rehabilitation has the following goals:

1. To validate a rehabilitation protocol in Immersive virtual reality (IVR) for restoring motor functions following peripheral injuries of the lower limbs. The protocol would be based on observation of actions rather than their execution. The rationale behind this idea is that indirect activation of the motor system through the observation of one's "own" virtual body that performs physical exercises would recruit the same neurocognitive mechanisms as those involved in the real motor control and action execution. This would improve the motor recovery by significantly enhancing the physical rehabilitation.
2. To develop a standard protocol that would combine the neuroscientific approach based on IVR and the standards of sport rehabilitation and would create a new approach that would complement the classical rehabilitation and could be executed remotely at home.

SAMPLE Participants will be recruited at HastaFisio and Centro di Medicina Preventiva e dello Sport dell'Università degli Studi di Torino physiotherapy center s; the sample will consist of adults (age range 18-65 years) that underwent knee sprain and/or surgery to knee ligaments and/or meniscus after musculoskeletal injuries of the knee. The sample size was estimated based on a priori power analysis for mixed-effects 3x3 ANOVA with Time (Pre, Mid, and Post) as within-subject factor and Group (Experimental, Active control, No VR) as between-subject factor. To reach a power of 0.80 with a medium effect size (f = 0.25) and alpha level set at 0.05, the required sample size is 36 (12 participants per group). The study will recruit 45 participants (15 per group) to account for possible dropouts.

METHODS The first experimental session will take place within two weeks from the knee surgery and the IVR training intervention will last six weeks, in parallel with the first phase of standard physical rehabilitation. The IVR training protocol implies observing a virtual avatar in the first-person perspective (Experimental group), or in the third-person perspective (Active control group); another control group (No IVR training) will undergo only the standard physical training. In the virtual scenario, the avatar will perform a series of rehabilitation exercises (see details below). Before (T0), in the middle (T1) and after (T2) the intervention, the neuromuscular functions will be assessed with a battery of standard clinical tests (see details below). Moreover, in order to evaluate the efficacy of the IVR procedure, embodiment will be measured via an ad hoc questionnaire at the same time points.

Measures:

The following battery of tests will be collected at T0, T1 and T2:

1. Before IVR training session:

   * IKDC scale (International knee documentation committee subjective knee evaluation form);
   * Joint position sense measured with GyKo (inertial measurement tool);
   * Knee extension range of motion measured with GyKo (inertial measurement tool);
   * Maximal force of the knee extensors measured via hand-held dynamometer;
   * Visual analogue scale (VAS) for pain after maximal contraction.
2. During the IVR training session:

   - Embodiment questionnaire after the exercises are completed.
3. After the IVR training session:

   * Subjective familiarity with each exercise presented in the IVR training;
   * General subjective feedback regarding the IVR session. Note that the clinical physiological measures (joint position sense, knee extension, maximal force of knee extensors) will be registered for both legs.

Training:

All groups of participants will follow two times per week the standard physical training protocol that will include exercises on strength, balance and flexibility. In addition, Experimental and Active control groups will participate in the IVR training administered on the same days as the physical training, always preceding it. The IVR training will be administered through a head-mounted display that allows presenting immersive 3D environments with a 360° field of view. The virtual scene will contain a gym with some standard equipment and a virtual avatar in natural size, gender-matched with the participants. The avatar will be seen either from the first-person perspective (i.e., as if the avatar replaced the real body; Experimental group), or from the third-person perspective (i.e., as if it was another person observed from the side; Active control group). After the initial familiarization and immersion phase, the avatar will perform a series of exercises (seated knee extension, squat, forward lunge, step up and down from a step, split squat, anterior reach of Y-balance test), 3 circuits with 8 repetition of each exercise, that imitate a real-life physical rehabilitation session. The avatar will perform the exercises on the injured-leg side (in cases when the exercises are one-legged).

Analysis:

The data obtained in the tests and questionnaires described above will be compared between the three groups (Experimental, Active control and No IVR training) and within the three time-points (T0, T1, T2) using a 3x3 mixed-effects ANOVA with Time as a within-subject factor and group as a between-subject factor. The hypothesis is that the Experimental group will show greater improvement in the injured limb's functional performance than the Active control group and No IVR training group.

IMPLICATIONS OF THE PROJECT From the theoretical perspective, the project will be the first to provide evidence of the fundamental role of the neurocognitive mechanisms underlying conscious representation of one's own body in motor rehabilitation of peripheral injuries. Indeed, at the present moment, only a few studies suggest that simply representing a body as one's own (without any need to perform movements) influences the motor system. Only one study examined whether this could have a positive influence on the motor functioning; however, those results were collected in patients with brain lesions, rather than peripheral ones. For these reasons, the project offers a new approach to rehabilitation that is based on hypothesis well-supported by the existing theoretical knowledge but remaining unexplored experimentally. Demonstrating that the illusion that one's own body was moving can promote the activation of brain areas involved in motor planning and execution (e.g., planning and execution of sport rehabilitation exercises), and therefore, improving the deficient motor functionality, would be a novel scientific finding. Moreover, demonstrating that the motor system can be affected through the signals related to the body via the properties of a virtual body, even in case of peripheral injuries, creates new opportunities in the more general context of motor rehabilitation.

In terms of impact on the rehabilitation science, the effects of the project outcomes will appear on several levels, since it proposes a radical change to the sport rehabilitation approach. The loss of motor functioning as a result of sport injuries is a debilitating event with a cascade of negative consequences. The state of the art of the rehabilitation includes standard protocols that are based on the execution of movements and that have to be performed in appropriately equipped structures (gyms of rehabilitation centers). Firstly, the IVR training does not require any physical movement execution, and therefore, can serve as a valuable addition to the standard rehabilitation protocols, or even replace some physical rehabilitation sessions. Secondly, IVR training can be performed remotely and autonomously by the patient, which is an important advantage for any type of intervention, especially in light of the current situation of the global pandemic. These two elements might greatly reduce the cumulative time and effort invested in the recovery from injuries. Thirdly, such approach is highly flexible by nature and can be complemented by other techniques and measures of motor behavior (e.g., movement kinematics, brain electrical activity, measures of the activity of the autonomic nervous system, etc.), depending on the specific needs and level of complexity.

ELIGIBILITY:
Inclusion Criteria:

* Early recovery after knee sprain and/or surgery to knee ligaments and/or meniscus after musculoskeletal injuries of the knee
* Normal or corrected-to-normal visual acuity

Exclusion Criteria:

* History of neurological or psychiatric disorders
* Motion sickness during IVR use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of the IKDC scale score from pre-training to post-training | T0 (Before VR training sessions), T1 (After 50% of VR training sessions, week 3), T2 (After 100% of VR training sessions, week 6)
  International knee documentation committee subjective knee evaluation form; scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Change of the joint position sense measure from pre-training to post-training | T0 (Before VR training sessions), T1 (After 50% of VR training sessions, week 3), T2 (After 100% of VR training sessions, week 6)
  Joint position sense measured with GyKo (inertial measurement tool)
Embodiment questionnaire pre-training | T0 (Before VR training sessions)
  Measure of subjective experience of body ownership/agency in the VR scenario on a visual analogue scale; min = 1, max = 10, where lower scores indicate absence of/weaker illusion of embodiment and higher scores indicate stronger illusion of embodiment
Embodiment questionnaire mid-training | T1 (After 50% of VR training sessions, week 3)
  Measure of subjective experience of body ownership/agency in the VR scenario on a visual analogue scale; min = 1, max = 10, where lower scores indicate absence of/weaker illusion of embodiment and higher scores indicate stronger illusion of embodiment
Embodiment questionnaire post-training | T2 (After 100% of VR training sessions, week 6)
  Measure of subjective experience of body ownership/agency in the VR scenario on a visual analogue scale; min = 1, max = 10, where lower scores indicate absence of/weaker illusion of embodiment and higher scores indicate stronger illusion of embodiment

SECONDARY OUTCOMES:
Change of the knee extension measure from pre-training to post-training | T0 (Before VR training sessions), T1 (After 50% of VR training sessions, week 3), T2 (After 100% of VR training sessions, week 6)
  Knee extension range of motion (degrees) measured with GyKo (inertial measurement tool)
Change of maximal force of the knee extensors from pre-training to post-training | T0 (Before VR training sessions), T1 (After 50% of VR training sessions, week 3), T2 (After 100% of VR training sessions, week 6)
  Maximal force of the knee extensors (N) measured via hand-held dynamometer
Change of subjective level of pain after maximal contraction from pre-training to post-training | T0 (Before VR training sessions), T1 (After 50% of VR training sessions, week 3), T2 (After 100% of VR training sessions, week 6)
  Subjective scale (visual analogue scale) for pain after maximal contraction of the knee; min score = 0, max score = 10, where lower scores indicate lower level of pain
Subjective feedback regarding the IVR experience pre-training | T0 (Before VR training sessions)
  Subjective familiarity with each exercise presented in the IVR training and general subjective feedback regarding the IVR session
Subjective feedback regarding the IVR experience mid-training | T1 (After 50% of VR training sessions, week 3)
  Subjective familiarity with each exercise presented in the IVR training and general subjective feedback regarding the IVR session
Subjective feedback regarding the IVR experience post-training | T2 (After 100% of VR training sessions, week 6)
  Subjective familiarity with each exercise presented in the IVR training and general subjective feedback regarding the IVR session

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Pia, PhD, Study Chair — University of Turin, Italy; Maria Pyasik, PhD, Principal Investigator — University of Turin, Italy; Gennaro Boccia, PhD, Principal Investigator — University of Turin, Italy
Locations (1):
- University of Turin, Turin, TO, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made publicly available in anonymized form via an online data repository (Mendeley data).
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available together with the publication of preprint/article reporting the results of the study.
Access Criteria: The data will be freely available.

REFERENCES:
- [Result] Burin D, Pyasik M, Salatino A, Pia L. That's my hand! Therefore, that's my willed action: How body ownership acts upon conscious awareness of willed actions. Cognition. 2017 Sep;166:164-173. doi: 10.1016/j.cognition.2017.05.035. Epub 2017 May 31. PMID 28577446
- [Result] Cumps E, Verhagen E, Annemans L, Meeusen R. Injury rate and socioeconomic costs resulting from sports injuries in Flanders: data derived from sports insurance statistics 2003. Br J Sports Med. 2008 Sep;42(9):767-72. doi: 10.1136/bjsm.2007.037937. Epub 2007 Nov 29. PMID 18048438
- [Result] Ekstrand J, Walden M, Hagglund M. Hamstring injuries have increased by 4% annually in men's professional football, since 2001: a 13-year longitudinal analysis of the UEFA Elite Club injury study. Br J Sports Med. 2016 Jun;50(12):731-7. doi: 10.1136/bjsports-2015-095359. Epub 2016 Jan 8. PMID 26746908
- [Result] Maselli A, Slater M. The building blocks of the full body ownership illusion. Front Hum Neurosci. 2013 Mar 21;7:83. doi: 10.3389/fnhum.2013.00083. eCollection 2013. PMID 23519597
- [Result] Pyasik M, Salatino A, Burin D, Berti A, Ricci R, Pia L. Shared neurocognitive mechanisms of attenuating self-touch and illusory self-touch. Soc Cogn Affect Neurosci. 2019 Feb 13;14(2):119-127. doi: 10.1093/scan/nsz002. PMID 30649514
- [Result] Pyasik M, Ronga I, Burin D, Salatino A, Sarasso P, Garbarini F, Ricci R, Pia L. I'm a believer: Illusory self-generated touch elicits sensory attenuation and somatosensory evoked potentials similar to the real self-touch. Neuroimage. 2021 Apr 1;229:117727. doi: 10.1016/j.neuroimage.2021.117727. Epub 2021 Jan 9. PMID 33434613
- [Result] Rossetti, Y., Rode, G., & Goldenberg, G. (2005). Perspectives in higher-order motor deficits rehabilitation: Which approach for which ecological result? In H. J. Freund, M. Jeannerod, M. Hallett, & R. Leiguarda (Eds.), Higher-order motor disorders: From neuroanatomy and neurobiology to clinical neurology (pp. 475-497). Oxford University Press.
- [Result] Tambone R, Giachero A, Calati M, Molo MT, Burin D, Pyasik M, Cabria F, Pia L. Using Body Ownership to Modulate the Motor System in Stroke Patients. Psychol Sci. 2021 May;32(5):655-667. doi: 10.1177/0956797620975774. Epub 2021 Apr 7. PMID 33826456
- [Result] Whatman C, Hing W, Hume P. Physiotherapist agreement when visually rating movement quality during lower extremity functional screening tests. Phys Ther Sport. 2012 May;13(2):87-96. doi: 10.1016/j.ptsp.2011.07.001. Epub 2011 Aug 27. PMID 22498149
- [Result] Winstein, C. J., & Wolf, S. L. (2008). Task-oriented training to promote upper extremity recovery. In J. Stein, R. Harvey, R. Macko, C. J. Winstein, & R. Zorowitz (Eds.), Stroke recovery and rehabilitation (pp. 267-290). Demos Medical Publishing.
- [Result] Pyasik M, Furlanetto T, Pia L. The Role of Body-Related Afferent Signals in Human Sense of Agency. J Exp Neurosci. 2019 May 16;13:1179069519849907. doi: 10.1177/1179069519849907. eCollection 2019. PMID 31205423